CLINICAL TRIAL: NCT00789633
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, 2-parallel Group, Phase III Study to Compare Efficacy and Safety of Masitinib 9 mg/kg/Day in Combination With Gemcitabine Compared to Placebo in Combination With Gemcitabine in Treatment of Patients With Advanced/Metastatic Pancreatic Cancer
Brief Title: Masitinib in Combination With Gemcitabine for Treatment of Patients With Advanced/Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB07012
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Advanced pancreatic cancer; Metastatic pancreatic cancer; Gemcitabine; Chemo-naive
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — masitinib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib & gemcitabine (Experimental): Participants receive masitinib (9 mg/kg/day), given orally twice daily, plus gemcitabine at 1000mg/m2 by intravenous infusion during 30 minutes, once every 7 days, for up to 7 weeks, followed by a week of rest. Subsequent cycles should consist of an IV infusion, once every 7 days, for 3 consecutive weeks out of every 4 weeks, until disease progression, death, limiting toxicity or patient consent withdrawal.
  Interventions: Drug: Masitinib; Drug: Gemcitabine
- Placebo & gemcitabine (Placebo Comparator): Participants receive matching placebo, given orally twice daily, plus gemcitabine at 1000mg/m2 by intravenous infusion during 30 minutes, once every 7 days, for up to 7 weeks, followed by a week of rest. Subsequent cycles should consist of an IV infusion, once every 7 days, for 3 consecutive weeks out of every 4 weeks, until disease progression, death, limiting toxicity or patient consent withdrawal.
  Interventions: Drug: Placebo; Drug: Gemcitabine

INTERVENTIONS:
Drug: Masitinib — Masitinib at 9 mg/kg/day given orally twice daily
  Other Names: AB1010
  Arms: Masitinib & gemcitabine
Drug: Placebo — Matching placebo given orally twice daily
  Arms: Placebo & gemcitabine
Drug: Gemcitabine — Gemcitabine at 1000 mg/m2 by intravenous infusion
  Other Names: Gemzar

SUMMARY:
The objective of this study is to compare the efficacy and safety of masitinib in combination with gemcitabine to placebo in combination with gemcitabine in patients with advanced/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Human pancreatic cancer overexpresses a number of important tyrosine kinase (TK) growth factors receptors and ligands, including expression of both PDGF and PDGF receptors. Drugs that can selectively inhibit TKs are likely to be of benefit in pancreatic cancer. Masitinib is a TK inhibitor, selectively and effectively inhibiting c-Kit (mast cell growth factor receptor), PDGF receptor, FGF receptor and to a lower extent the FAK kinases. Pre-clinical and clinical studies have shown that masitinib can reverse resistance of pancreatic tumor cell lines to gemcitabine. Based on pre-clinical and phase 2 clinical studies, masitinib can be considered as a good candidate to use in combination with gemcitabine in the treatment of pancreatic cancer.

ELIGIBILITY:
Main Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas
2. Chemo naïve patients with advanced/metastatic disease
3. Documented decision justifying non eligibility for surgical resection. The documentation of the non eligibility for surgical resection will be reviewed by an independent committee.
4. Men and women, age >18 years
5. Men and women of childbearing potential (entering the study after a confirmed menstrual period and who have a negative pregnancy test), must agree to use two methods (one for the patient and one for the partner) of medically acceptable forms of contraception during the study and for 3 months after the last treatment intake.
6. Patient should be able and willing to comply with study visits and procedures as per protocol.
7. Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.

Main Exclusion Criteria:

1. Patient treated for a cancer other than pancreatic cancer within 5 years before enrollment, with the exception of basal cell carcinoma or in situ cervical cancer
2. Any condition that the physician judges could be detrimental to subjects participating in this study; including any clinically important deviations from normal clinical laboratory values or concurrent medical events Previous treatment
3. Any anti-tumor therapy (any chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy) within 6 months prior to baseline
4. Treatment with any investigational agent within 4 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2008-11-25 (Actual); Primary Completion 2011-12-23 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From day of randomization to the date of death, assessed up to 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Survival rate | Every 24 weeks, assessed up to 60 months
  Defined as the proportion of patients alive at each time point, estimated with Kaplan-Meier distribution.
Progression Free Survival (PFS) | From day of randomization to disease progression or death, whichever came first, assessed up to 60 months
  Progression Free Survival is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by the investigator on CT scan according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gaël Deplanque, MD, Principal Investigator — Hôpital Saint Joseph, Paris, France
Locations (67):
- United States (12):
  - Eastern Connecticut Hematology and Oncology (ECHO), Norwich, Connecticut
  - MD Anderson, Orlando, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - Medical & Surgical Specialists, Galesburg, Illinois
  - Berkshire Hematology Oncology, Pittsfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Metro MN CCOP, Saint Louis Park, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - The Valley Hospital, Paramus, New Jersey
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oregon Health & Science University, Portland, Oregon
- Czechia (7):
  - Teaching Hospital Brno-Bohunice, Brno
  - Hospital Chomutov, Chomutov
  - Oncology Surgery, Kutná Hora
  - Department of Oncology Teaching Hospital Olomouc, Olomouc
  - Teaching Hospital Královské, Prague
  - Teaching Hospital Na Bulovce, Prague
  - Hospital na Homolce, Prague
- France (36):
  - CHU Amiens, Amiens
  - Hôpital Privé d'Antony, Antony
  - Institut Sainte-Catherine, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Saint-André, Bordeaux
  - CHU de la Cavale Blanche, Brest
  - CHU de Caen, Caen
  - CHU Hôtel Dieu, Clermont-Ferrand
  - Groupement Hospitalier Universitaire Nord - Beaujon, Clichy
  - CHU Henri Mondor, Créteil
  - Hôpital Victor Jousselin, Dreux
  - Centre Gastro-Loire, Gien
  - Institut Daniel Hollard, Grenoble
  - CHD Les Oudairies, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Robert Boulin, Libourne
  - Hôpital Claude Huriez, Lille
  - Centre Hospitalier de Longjumeau, Longjumeau
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Centre Léon Bérard, Lyon
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Hôpital Saint Joseph, Marseille
  - Centre Hospitalier Belfort - Montbéliard, Montbéliard
  - CHU Hôtel Dieu, Nantes
  - Centre Catherine de Sienne, Nantes
  - Hôpital de la Source, Orléans
  - Groupe Hospitalier Diaconesse Croix Saint Simon, Paris
  - Hôpital Tenon, Paris
  - Hôpital Hôtel Dieu, Paris
  - Hôpital Saint-Joseph, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Polyclinique Francheville, Périgueux
  - Hôpital Hautepierre, Strasbourg
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif
- Lebanon (7):
  - Hotel Dieu de France, Beirut
  - Makassed General Hospital Tarik Jadide, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Saint Georges Hospital UMC, Beirut
  - Middle East Institute of Health- Bsaleem, Metn
  - Saint Joseph Hospital Baouchrieh, Metn
  - Hammoud Hospital University Medical Center, Saida
- Romania (5):
  - Municipal Clinical Hospital, Arad
  - County Hospital, Baia Mare
  - Emergency Clinical Hospital, Constanța
  - Pelica Impex SRL Hospital, Pelica Impex
  - County Hospital, Satu Mare

REFERENCES:
- [Result] Deplanque G, Demarchi M, Hebbar M, Flynn P, Melichar B, Atkins J, Nowara E, Moye L, Piquemal D, Ritter D, Dubreuil P, Mansfield CD, Acin Y, Moussy A, Hermine O, Hammel P. A randomized, placebo-controlled phase III trial of masitinib plus gemcitabine in the treatment of advanced pancreatic cancer. Ann Oncol. 2015 Jun;26(6):1194-1200. doi: 10.1093/annonc/mdv133. Epub 2015 Apr 9. PMID 25858497
- See also: Link to article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4516046/